CLINICAL TRIAL: NCT05906771
Title: Study of the Effect of the Combined Extract of Lemon Verbena and Hibiscus on Health Indicators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alicante (Other)
Responsible Party: Principal Investigator, Prof. Dr. Alejandro Martínez-Rodríguez, Full Professor, University of Alicante
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UA-2023-05-08
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Diet, Mediterranean; Antioxidant Effect; Body Weight; Cardiovascular Diseases; Densitometry; Body Composition
MeSH Terms: conditions — Body Weight; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP (Placebo Comparator): Nutraceutical placebo intake group
  Interventions: Dietary Supplement: Nutraceutical placebo
- EXPERIMENTAL GROUP (Experimental): Intake of natural herbal dietary supplement composed of a combination of Hibiscus sabdariffa flowers and Lippia citriodora leaves.
  Interventions: Dietary Supplement: Metabolaid(R)

INTERVENTIONS:
Dietary Supplement: Metabolaid(R) — The participating subjects will have to follow the intake of the nutraceutical for 3 months, as well as attend the stipulated visits. Participants will be given a register to control their daily intake of the nutraceutical. They should not change their daily habits.
  The nutraceutical has been elaborated by Monteloeder, S.L. It is a combination of Hibiscus sabdariffa flowers and Lippia citriodora leaves. The dose that the participants of the experimental group will receive will be 300mg plus 20mg of microcrystalline cellulose. The product is presented in an unflavored capsule, it is a reddish-brown powder with a characteristic odor and a slightly bitter taste. The manufacturing date of the product was 01/12/2022 and the expiration date was 30/11/2024.
  Arms: EXPERIMENTAL GROUP
Dietary Supplement: Nutraceutical placebo — The participating subjects will have to follow the intake of the nutraceutical for 3 months, as well as attend the stipulated visits. Participants will be given a register to control their daily intake of the nutraceutical. They should not change their daily habits.
  Nutraceutical placebo contains microcystalline cellulose (185mg) and maltodextrin (185mg).
  Arms: CONTROL GROUP

SUMMARY:
Plant polyphenols have demonstrated the ability to ameliorate metabolic alterations induced by overweight and obesity, both in cellular and animal models, where most therapeutic approaches have failed. These have demonstrated the ability to improve appetite sensation, leading to improved body weight control, in addition to reducing fat accumulation and improving plasma glycemic and lipid profiles, as well as inflammatory process and vascular dysfunction. The plant polyphenols on which the extract to be studied will be based will be hibiscus and lemon verbena. A randomized controlled trial will be carried out in overweight or obese subjects from the province of Alicante. An electronic randomization will be carried out based on a two-branch design, therefore, there will be a control group (no intervention) and an experimental group (nutraceutical intake). Participants will have to ingest the nutraceutical for 3 months, as well as attend the agreed visits. Different satiety questionnaires, circulating parameters measured in capillaries (cholesterol, triglycerides and glucose), blood pressure and body composition measured by bone densitometry (DXA) will be collected. All variables will be measured at 4 different time points (baseline, 30 days, 60 days and 90 days). All these will be analyzed as a function of time; at the beginning and end of each intervention (intra-group analysis), as well as comparing the control group with the experimental group (inter-group analysis). A multidisciplinary team formed by physicians, nurses and nutritionists will be involved.

ELIGIBILITY:
Inclusion Criteria:

* Elderly (< 18 years)
* Overweight (body mass index 25-29.9 kg/m2)

Exclusion Criteria:

* Pregnant or lactating subjects
* Who have participated in another study with similar characteristics in the last 3 months.
* Subjects with pathologies.
* Consumption of drugs and/or supplements
* Subjects with food intolerances/allergies.
* Subjects with muscle or joint injury.
* Subjects with impossibility to follow up the intervention.
* Refusal of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
WEIGHT | 12 weeks
  The weight of the subjects will be obtained using the TANITA (Tokyo, Japan).
HEIGHT | 12 weeks
  The height of the subjects will be measured with the SECA 123 stadiometer (Hamburg, Germany).
BLOOD PREASURE | 12 weeks
  Measurement of blood pressure (systolic and diastolic) with a digital tensiometer.
FAT MASS | 12 weeks
  Assessment of body composition by DXA and bioimpedance to obtain fat mass results.
HEART RATE | 12 weeks
  Measurement of heart rate with a digital tensiometer.
SATIETY | 12 weeks
  Scores will be obtained through validated questionnaires for the study of satiety of the participating subjects.
BLOOD CHOLESTEROL LEVEL | 12 weeks
  Cholesterol blood values will be obtained using the flexible and portable accutrend® plus
TRIGLICERIDES | 12 weeks
  Triglicerides blood values will be obtained using the flexible and portable accutrend® plus
BLOOD GLUCOSE LEVEL | 12 weeks
  Glucose blood values will be obtained using the flexible and portable accutrend® plus

CONTACTS AND LOCATIONS:
Locations (1):
- Alejandro Martínez Rodríguez, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No